CLINICAL TRIAL: NCT00003805
Title: Vancomycin Versus Placebo in Persistently Febrile Granulocytopenic Patients Given Piperacillin/Tazobactam
Brief Title: Prevention of Infection in Patients With Hematologic Cancer and Persistent Fever Caused by a Low White Blood Cell Count
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Supportive Care
Other Study IDs: EORTC-46971; EORTC-46971
Record Dates: First submitted 1999-11-01; First posted 2004-07-16 (Estimated); Last update posted 2012-09-24 (Estimated); Status verified 2012-09

CONDITIONS: Bone Marrow Suppression; Fever, Sweats, and Hot Flashes; Infection; Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes; Unspecified Adult Solid Tumor, Protocol Specific; Unspecified Childhood Solid Tumor, Protocol Specific
Keywords: stage I adult Hodgkin lymphoma; stage II adult Hodgkin lymphoma; stage III adult Hodgkin lymphoma; stage IV adult Hodgkin lymphoma; recurrent childhood acute lymphoblastic leukemia; recurrent adult Hodgkin lymphoma; stage I cutaneous T-cell non-Hodgkin lymphoma; stage II cutaneous T-cell non-Hodgkin lymphoma; stage III cutaneous T-cell non-Hodgkin lymphoma; stage IV cutaneous T-cell non-Hodgkin lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; Burkitt lymphoma; stage 0 chronic lymphocytic leukemia; Waldenstrom macroglobulinemia; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; stage I childhood lymphoblastic lymphoma; stage II childhood lymphoblastic lymphoma; stage III childhood lymphoblastic lymphoma; stage IV childhood lymphoblastic lymphoma; recurrent childhood lymphoblastic lymphoma; stage I chronic lymphocytic leukemia; stage II chronic lymphocytic leukemia; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; recurrent childhood acute myeloid leukemia; recurrent adult acute myeloid leukemia; recurrent adult acute lymphoblastic leukemia; relapsing chronic myelogenous leukemia; refractory chronic lymphocytic leukemia; childhood diffuse large cell lymphoma; childhood immunoblastic large cell lymphoma; unspecified childhood solid tumor, protocol specific; unspecified adult solid tumor, protocol specific; chronic phase chronic myelogenous leukemia; accelerated phase chronic myelogenous leukemia; blastic phase chronic myelogenous leukemia; meningeal chronic myelogenous leukemia; adult acute myeloid leukemia in remission; adult acute lymphoblastic leukemia in remission; childhood acute myeloid leukemia in remission; childhood acute lymphoblastic leukemia in remission; fever, sweats, and hot flashes; progressive hairy cell leukemia, initial treatment; refractory hairy cell leukemia; stage II childhood Hodgkin lymphoma; stage I childhood Hodgkin lymphoma; stage III childhood Hodgkin lymphoma; stage IV childhood Hodgkin lymphoma; recurrent/refractory childhood Hodgkin lymphoma; stage I grade 2 follicular lymphoma; stage I grade 3 follicular lymphoma; stage I adult diffuse small cleaved cell lymphoma; stage I adult diffuse mixed cell lymphoma; stage I adult diffuse large cell lymphoma; stage I adult immunoblastic large cell lymphoma; stage I adult lymphoblastic lymphoma; stage I adult Burkitt lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse large cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III adult Burkitt lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV adult Burkitt lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; stage I adult T-cell leukemia/lymphoma; stage II adult T-cell leukemia/lymphoma; stage III adult T-cell leukemia/lymphoma; stage IV adult T-cell leukemia/lymphoma; recurrent adult T-cell leukemia/lymphoma; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; infection; bone marrow suppression; stage I childhood small noncleaved cell lymphoma; stage I childhood large cell lymphoma; stage II childhood small noncleaved cell lymphoma; stage II childhood large cell lymphoma; stage III childhood small noncleaved cell lymphoma; stage III childhood large cell lymphoma; stage IV childhood small noncleaved cell lymphoma; stage IV childhood large cell lymphoma; recurrent childhood small noncleaved cell lymphoma; recurrent childhood large cell lymphoma; stage I mantle cell lymphoma; contiguous stage II grade 1 follicular lymphoma; contiguous stage II grade 2 follicular lymphoma; contiguous stage II grade 3 follicular lymphoma; contiguous stage II adult diffuse small cleaved cell lymphoma; contiguous stage II mantle cell lymphoma; contiguous stage II adult diffuse mixed cell lymphoma; contiguous stage II adult immunoblastic large cell lymphoma; contiguous stage II adult diffuse large cell lymphoma; contiguous stage II adult Burkitt lymphoma; contiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II mantle cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma; recurrent mantle cell lymphoma; contiguous stage II marginal zone lymphoma; contiguous stage II small lymphocytic lymphoma; noncontiguous stage II small lymphocytic lymphoma; noncontiguous stage II marginal zone lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; stage I marginal zone lymphoma; stage I small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage III marginal zone lymphoma; stage IV small lymphocytic lymphoma; stage IV marginal zone lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; childhood myelodysplastic syndromes
MeSH Terms: conditions — Fever; Hot Flashes; Infections; Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Hodgkin Disease; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, T-Cell, Cutaneous; Burkitt Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Waldenstrom Macroglobulinemia; Leukemia, Myeloid, Acute; Lymphoma, Large B-Cell, Diffuse; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myeloid, Accelerated Phase; Blast Crisis; Leukemia, Hairy Cell; Recurrence; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Dendritic Cell Sarcoma, Interdigitating; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone | interventions — Piperacillin; Piperacillin, Tazobactam Drug Combination; Tazobactam; Vancomycin

INTERVENTIONS:
Drug: piperacillin sodium
Drug: piperacillin-tazobactam
Drug: tazobactam sodium
Drug: vancomycin

SUMMARY:
RATIONALE: Antibiotic therapy may prevent the development of infection in patients with hematologic cancer and the persistent fever caused by a low white blood cell count. It is not yet known which regimen of antibiotics is most effective in preventing infection in these patients.

PURPOSE: Randomized phase III trial to study the effectiveness of piperacillin-tazobactam with or without vancomycin in reducing fever in patients who have leukemia, lymphoma, or Hodgkin's disease.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the efficacy of piperacillin and tazobactam with or without vancomycin in reducing fever in patients with hematological malignancies and persistent febrile granulocytopenia.

OUTLINE: This is a randomized, double blind, multicenter study. Patients receive piperacillin/tazobactam IV over 20-30 minutes every 6 hours. Patients who become afebrile within 48-60 hours after beginning treatment continue to receive piperacillin/tazobactam alone. These afebrile patients continue treatment for a minimum of 7 days, of which 4 must be consecutive without fever. Patients who are still febrile after the initial 48-60 hours are randomized to continue on piperacillin/tazobactam alone or with vancomycin. Vancomycin IV is administered over at least 1 hour twice daily. Treatment continues for a maximum of 28 days in the absence of persistent fever. Patients are followed at 7-10 days after completion of therapy.

PROJECTED ACCRUAL: A total of 500 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Leukemia, lymphoma, or Hodgkin's disease OR Stem cell transplantation or bone marrow transplantation (allogenic or autologous) for a neoplastic disease Absolute granulocyte count no greater than 1,000/mm3 anticipated to fall below 500/mm3 within 24-48 hours, and expected to last for longer than 7 days from onset of fever Fever (i.e., oral or axillary temperature at least 38.5 degrees C or 101.3 degrees F once, or at least 38 degrees C or 100.4 degrees F on two or more occasions separated at least by 1 hour during a 12 hour period) Presumed infection

PATIENT CHARACTERISTICS: Age: 2 and over Performance status: Not moribund or comatose for any reason with little hope of recovery Life expectancy: At least 48 hours Hematopoietic: See Disease Characteristics Hepatic: No hepatic stupor or coma Renal: Adults: No renal failure requiring hemodialysis or peritoneal dialysis OR Creatinine no greater than 2.25 mg/dL OR Creatinine clearance at least 40 mL/min Children: No renal impairment (i.e., creatinine greater than upper limit of normal) Pulmonary: No lung infiltrate Other: No known allergy to piperacillin, tazobactam, or vancomycin No history of immediate or accelerated reaction to beta-lactam antibiotics No prior inclusion in this study No catheter related infection No known HIV infection Not pregnant or nursing

PRIOR CONCURRENT THERAPY: Biologic therapy: See Disease Characteristics Chemotherapy: Not specified Endocrine therapy: Not specified Radiotherapy: Not specified Surgery: Not specified Other: At least 4 days since prior intravenous antibacterial agents Oral antibiotics for prophylaxis of bacterial infection allowed At least 30 days since prior treatment with any other investigational antibiotic No other concurrent antibiotics except trimethoprim-sulfamethoxazole for the prevention of Pneumocystis carinii pneumonia

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 859 (Actual)
Dates: Start 1997-11; Primary Completion 2000-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michel P. Glauser, MD, Study Chair — Centre Hospitalier Universitaire Vaudois
Locations (28):
- United States (2):
  - Marlene & Stewart Greenebaum Cancer Center, University of Maryland, Baltimore, Maryland
  - Boston Medical Center, Boston, Massachusetts
- Belgium (4):
  - Algemeen Ziekenhuis Middelheim, Antwerp
  - Hopital Universitaire Erasme, Brussels
  - Institut Jules Bordet, Brussels (Bruxelles)
  - Cliniques Universitaires Saint-Luc, Brussels (Bruxelles)
- Canada (2):
  - Kingston General Hospital, Kingston, Ontario
  - Ottawa Regional Cancer Center - General Division, Ottawa, Ontario
- Masaryk University Hospital, Brno, Czechia
- Turku University Central Hospital, Turku, Finland
- CHR de Besancon - Hopital Saint-Jacques, Besançon, France
- Klinikum der Universitaet Ulm, Ulm, Germany
- Greece (4):
  - Hellenic Institute for Cancer-Saint Savas Hospital, Athens
  - Athens University-Laikon General Hospital, Athens
  - Metaxa's Memorial Cancer Hospital, Piraeus
  - University of Patras Medical School, Rio Patras
- Israel (3):
  - Wolfson Medical Center, Holon
  - Hadassah University Hospital, Jerusalem
  - Chaim Sheba Medical Center, Ramat Gan
- Slovakia (2):
  - National Cancer Institute - Bratislava, Bratislava
  - St. Elizabeth Cancer Institute Hospital, Bratislava
- Switzerland (3):
  - Ospedale San Giovanni, Bellinzona
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - Universitaetsspital, Zurich
- Turkey (Türkiye) (3):
  - Ibn-i Sina Hospital, Ankara Univeristy, Ankara
  - Section of Infectious Diseases, Ankara
  - Marmara University Hospital, Istanbul
- Royal Marsden Hospital, Sutton, England, United Kingdom